CLINICAL TRIAL: NCT03662022
Title: Post ExpOsure Prophylaxis for LEprosy in the Comoros and Madagascar
Acronym: PEOPLE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: Damien Foundation (Other); Centre d'Infectiologie Charles Mérieux (Other); Fondation Raoul Follereau (Unknown); Leiden University Medical Center (Other); L'Institut National de la Santé et de la Recherche Médicale (Unknown); Genoscreen (Other); Instituto Fernandes Figueira (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1248/18
Record Dates: First submitted 2018-09-05; First posted 2018-09-07 (Actual); Results first posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Leprosy
MeSH Terms: conditions — Leprosy | interventions — Rifampin

STUDY DESIGN:
Intervention Model Description: A cluster randomized trial in which villages are assigned to one of four intervention groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- No PEP (No Intervention): No PEP will be distributed
- Household PEP (Other): PEP will be given to all household contacts of an incident leprosy patient
  Interventions: Drug: Rifampicin
- PEP 100m (Experimental): PEP will be given to all household contacts of leprosy patients and to all other people living within a 100m radius of an incident leprosy patient.
  Interventions: Drug: Rifampicin
- PEP 100m + positive for anti-PGL-I IgM Ab (Other): PEP will be given to all household contacts of leprosy patients and to all other people living within a 100m radius of an incident leprosy patient who test positive in the UCP-LFA detecting anti-M. leprae PGL-I IgM Ab in fingerstick blood (anti-PGL-I)
  Interventions: Drug: Rifampicin

INTERVENTIONS:
Drug: Rifampicin — Rifampicin will be given in the same way to arms 2, 3 and 4 (weight dependent). Only the strategy of whom to offer PEP differs between the arms.
  Arms: Household PEP; PEP 100m; PEP 100m + positive for anti-PGL-I IgM Ab

SUMMARY:
This is a cluster randomized trial on effectiveness of different modalities of Single Double Dose of Rifampicin Post-Exposure Prophylaxis (SDDR-PEP) for leprosy in the Comoros (Anjouan and Mohéli) and Madagascar.

The study aims to identify which approach to the selection of contacts for post exposure prophylaxis is most effective to reduce incident leprosy, and to Interrupt ongoing transmission from asymptomatic persons in the process of developing multibacillary leprosy.

DETAILED DESCRIPTION:
For the purpose of the study, villages on the Comoros and Madagascar that will be randomly assigned to one of the study arms, will be screened on a yearly basis for 4 consecutive years. Depending on which of the 4 arms a village is assigned to, people in the surroundings of a leprosy patient will or will not be offered Post-Exposure Prophylaxis (PEP) using rifampicin at 20mg/kg single dose:

1. No Post-Exposure Prophylaxis (PEP) is given to anyone
2. PEP is given to all household contacts of incident leprosy cases
3. PEP is given to all people who live in a 100m radius of incident leprosy cases
4. PEP is given to all household contacts of incident leprosy cases as well as to all others who live within a 100m radius of an incident leprosy case and test positive in the UCP-LFA detecting anti-M. leprae PGL-I IgM antibodies (Ab) in fingerstick blood (anti-PGL-1)

ELIGIBILITY:
Inclusion Criteria:

* Living in one of the study villages
* Aged 2 years and above
* Able and willing to provide informed consent

Exclusion Criteria:

* Signs of active leprosy (*)
* Signs of active pulmonary tuberculosis (cough ≥2 weeks duration) (*)
* Having received Rifampicin within the last 24 months (*)

(*) These people may still be included for yearly leprosy screening, but will be excluded to receive PEP

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 144000 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2023-01-17 (Actual); Study Completion 2023-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bouke de Jong, MD, PhD, Study Chair — Institute of Tropical Medicine; Epco Hasker, MD, Study Director — Institute of Tropical Medicine; Younoussa Assoumani, MD, Principal Investigator — Damien Foundation; Bertrand Cauchoix, MD, Principal Investigator — Fondation Raoul Follereau
Locations (3):
- Comoros (2):
  - Damien Foundation, Anjouan
  - Damien Foundation, Mohéli
- Fondation Raoul Follereau, Miandrivazo, Menabe Region, Madagascar

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Hasker E, Assoumani Y, Randrianantoandro A, Ramboarina S, Braet SM, Cauchoix B, Baco A, Mzembaba A, Salim Z, Amidy M, Grillone S, Attoumani N, Grillone SH, Ronse M, Peeters Grietens K, Rakoto-Andrianarivelo M, Harinjatovo H, Supply P, Snijders R, Hoof C, Tsoumanis A, Suffys P, Rasamoelina T, Corstjens P, Ortuno-Gutierrez N, Geluk A, Cambau E, de Jong BC. Post-exposure prophylaxis in leprosy (PEOPLE): a cluster randomised trial. Lancet Glob Health. 2024 Jun;12(6):e1017-e1026. doi: 10.1016/S2214-109X(24)00062-7. PMID 38762282
- [Derived] Marijke Braet S, Jouet A, Aubry A, Van Dyck-Lippens M, Lenoir E, Assoumani Y, Baco A, Mzembaba A, Cambau E, Vasconcellos SEG, Rigouts L, Suffys PN, Hasker E, Supply P, de Jong BC. Investigating drug resistance of Mycobacterium leprae in the Comoros: an observational deep-sequencing study. Lancet Microbe. 2022 Sep;3(9):e693-e700. doi: 10.1016/S2666-5247(22)00117-3. Epub 2022 Jul 15. PMID 35850123
- [Derived] Ortuno-Gutierrez N, Younoussa A, Randrianantoandro A, Braet S, Cauchoix B, Ramboarina S, Baco A, Mzembaba A, Salim Z, Amidy M, Grillone S, Richardus JH, de Jong BC, Hasker E. Protocol, rationale and design of PEOPLE (Post ExpOsure Prophylaxis for LEprosy in the Comoros and Madagascar): a cluster randomized trial on effectiveness of different modalities of implementation of post-exposure prophylaxis of leprosy contacts. BMC Infect Dis. 2019 Dec 5;19(1):1033. doi: 10.1186/s12879-019-4649-0. PMID 31805862

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Some participants will not have been present during the door to door screening of each year. It is possible that some pts will only have been screened in a limited number of periods. This explains the discrepancy between the enrollment nr in the protocol section and the pts assigned to the arms in period 1 (and other periods).Please note that the pts counts in the 'baseline characteristics' are the total of all started pts (in all years). This number reflects the total number analyzed.
Units Other Than Participants: Villages
Period: Year 1 2019
Arm/Group | No PEP | Household PEP | PEP 100m | PEP 100m + Positive for Anti-PGL-I IgM Ab
Started (participants examined) | 24185; 8 Villages | 23572; 8 Villages | 27196; 8 Villages | 19174; 8 Villages
Completed (participants under follow up) | 24102; 8 Villages | 23456; 8 Villages | 27038; 8 Villages | 19075; 8 Villages
Not Completed | 83; 0 Villages | 116; 0 Villages | 158; 0 Villages | 99; 0 Villages
Not completed — prevalent case | 83 | 116 | 158 | 99
Period: Year 2 2020
Arm/Group | No PEP | Household PEP | PEP 100m | PEP 100m + Positive for Anti-PGL-I IgM Ab
Started (under follow up from last year + examined for first time) | 25588; 8 Villages | 25419; 8 Villages | 28430; 8 Villages | 20910; 8 Villages
Completed (participants under follow up) | 23919; 8 Villages | 24202; 8 Villages | 27017; 8 Villages | 18002; 8 Villages
Not Completed | 1669; 0 Villages | 1217; 0 Villages | 1413; 0 Villages | 2908; 0 Villages
Not completed — incident case | 18 | 18 | 16 | 26
Not completed — other case | 18 | 16 | 16 | 24
Not completed — Lost to Follow-up | 1633 | 1183 | 1381 | 2858
Period: Year 3 2021
Arm/Group | No PEP | Household PEP | PEP 100m | PEP 100m + Positive for Anti-PGL-I IgM Ab
Started (under follow up from last year + examined for first time) | 24893; 8 Villages | 25257; 8 Villages | 28175; 8 Villages | 19511; 8 Villages
Completed (participants under follow up) | 24686; 8 Villages | 24971; 8 Villages | 27661; 8 Villages | 19009; 8 Villages
Not Completed | 207; 0 Villages | 286; 0 Villages | 514; 0 Villages | 502; 0 Villages
Not completed — incident case | 24 | 27 | 24 | 11
Not completed — other case | 4 | 15 | 10 | 14
Not completed — Lost to Follow-up | 179 | 244 | 480 | 477
Period: Year 4 2022
Arm/Group | No PEP | Household PEP | PEP 100m | PEP 100m + Positive for Anti-PGL-I IgM Ab
Started (under follow up from last year + examined for first time) | 25431; 8 Villages | 25760; 8 Villages | 28468; 8 Villages | 20605; 8 Villages
Completed (participants under follow up) | 24412; 8 Villages | 24621; 8 Villages | 27191; 8 Villages | 18765; 8 Villages
Not Completed | 1019; 0 Villages | 1139; 0 Villages | 1277; 0 Villages | 1840; 0 Villages
Not completed — incident case | 25 | 41 | 28 | 7
Not completed — other case | 8 | 19 | 13 | 7
Not completed — Lost to Follow-up | 986 | 1079 | 1236 | 1826

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No PEP | Household PEP | PEP 100m | PEP 100m + Positive for Anti-PGL-I IgM Ab | Total
Number analyzed (Participants) | 27494 | 27519 | 30709 | 24944 | 110666
Age, Customized [Count of Participants; unit: Participants] — Population: number analyzed in row differs from overall due to missing information
  Participants
    <5 years old: number analyzed (Participants) | 4509 | 4742 | 5257 | 4018 | 18526
    <5 years old | 4509 | 4742 | 5257 | 4018 | 18526
    =>5 and <15 years old: number analyzed (Participants) | 7775 | 8192 | 9062 | 7455 | 32484
    =>5 and <15 years old | 7775 | 8192 | 9062 | 7455 | 32484
    >=15 and <25 years old: number analyzed (Participants) | 5483 | 5300 | 6233 | 5001 | 22017
    >=15 and <25 years old | 5483 | 5300 | 6233 | 5001 | 22017
    25 years old and up: number analyzed (Participants) | 9722 | 9283 | 10156 | 8464 | 37625
    25 years old and up | 9722 | 9283 | 10156 | 8464 | 37625
    Missing: number analyzed (Participants) | 5 | 2 | 1 | 6 | 14
    Missing | 5 | 2 | 1 | 6 | 14
Sex: Female, Male [Count of Participants; unit: Participants] — Population: For both the second and fourth arm, there was one participant for which sex was missing
  Participants
    number analyzed (Participants) | 27494 | 27518 | 30709 | 24943 | 110664
    Female | 13978 | 13804 | 15303 | 12740 | 55825
    Male | 13516 | 13714 | 15406 | 12203 | 54839
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 27494 | 27519 | 30709 | 24944 | 110666
Region of Enrollment [Count of Participants; unit: Participants] — Population: numer analyzed in row differs form overall because of missing data.
  Participants
    Madagascar: number analyzed (Participants) | 4753 | 7087 | 5244 | 4074 | 21158
    Madagascar | 4753 | 7087 | 5244 | 4074 | 21158
    Comoros: number analyzed (Participants) | 22741 | 20432 | 25465 | 20870 | 89508
    Comoros | 22741 | 20432 | 25465 | 20870 | 89508
BCG scar [Count of Participants; unit: Participants]
  absent | 7886 | 8632 | 11897 | 11027 | 39442
  present | 18796 | 17960 | 17919 | 12585 | 67260
  missing | 812 | 926 | 893 | 1331 | 3962
Prevalent case [Count of Participants; unit: Participants] | 83 | 116 | 158 | 99 | 456
incident case [Count of Participants; unit: Participants] | 67 | 86 | 68 | 44 | 265
other case [Count of Participants; unit: Participants] | 30 | 50 | 39 | 45 | 164
receive PEP but ineligible or were elibile but did not receive PEP [Count of Participants; unit: Participants] | 0 | 155 | 5123 | 1336 | 6614

OUTCOME MEASURES:

1. Primary Outcome: Compare Effectiveness in Curbing Transmission of Leprosy of Three Different Approaches of Post Exposure Prophylaxis
Description: leprosy number of new cases per 1000 person years is reported. Incident cases were cases newly diagnosed while under follow-up.
  In the statisical analysis table: three incidence rate ratios between the comparator arm (arm 1) and each of the three intervention arms. These ratios will be based on incidence rates measured between the first and fourth household survey in each of the intervention arms, always divided by that of the comparator arm.
  Please note that accross the years a part of the same participants are revisited again, which might explain discrepancies in the overall number of participants analyzed.
Time Frame: 45 months
Population: participants examined
Measure: Number (95% Confidence Interval); unit: number of new cases per 1000 person/year
Groups:
- no PEP: no PEP given
Arm/Group | no PEP | Household PEP | PEP 100m | PEP 100m + Positive for Anti-PGL-I IgM Ab
Number analyzed (Participants) | 27494 | 27519 | 30709 | 24944
number of new cases per 1000 person/year | 1.04 [0.8 to 1.32] | 1.42 [1.13 to 1.75] | 0.98 [0.76 to 1.24] | 0.92 [0.67 to 1.23]
Statistical Analysis 1: Comparison: no PEP vs Household PEP; Test type: Superiority; p < 0.017, Mixed Models Analysis — The significance level was determined at 0.017, to account for the fact that we made three comparisons, thus conclusions can be drawn by examining if the 98.3% CI for the incidence rate ratio (IRR) contains the critical value of 1; incidence rate ratio = 0.95, 98.3% CI 2-sided [0.40 to 2.23]
Statistical Analysis 2: Comparison: no PEP vs PEP 100m; Test type: Superiority; p = 0.017, Mixed Models Analysis; incidence rate ratio = 0.80, 98.3% CI 2-sided [0.34 to 1.87]
Statistical Analysis 3: Comparison: no PEP vs PEP 100m + Positive for Anti-PGL-I IgM Ab; Test type: Superiority; p < 0.017, Mixed Models Analysis; incidence rate ratio = 0.58, 98.3% CI 2-sided [0.22 to 1.56]

ADVERSE EVENTS:
Time Frame: 1 day (during PEP administration visit) per year. Throughout the study (4 years) passive reporting was possible.
Description: There have been no adverse Events reported until now. Participants have been invited to report any adverse events to the study teams while they are present in the villages, the median duration the teams were present in a village in 2022 for example was 20 days. However no such events have been reported.
  For the no PEP arm, no adverse events were monitored/assessed.
Arm/Group | No PEP | Household PEP | PEP 100m | PEP 100m + Positive for Anti-PGL-I IgM Ab
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/731 | 0/15203 | 0/2850
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/731 | 0/15203 | 0/2850
Other Adverse Events (participants affected / at risk) | 0/0 | 0/731 | 0/15203 | 0/2850

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-03-18): https://cdn.clinicaltrials.gov/large-docs/22/NCT03662022/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-24): https://cdn.clinicaltrials.gov/large-docs/22/NCT03662022/SAP_001.pdf